CLINICAL TRIAL: NCT03466073
Title: A Double-blind, Placebo-controlled, Dose-escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Recombinant Human Plasma Gelsolin Added to Standard of Care in Subjects Hospitalized for Acute Community-acquired Pneumonia
Brief Title: A Phase 1b/2a Study of the Safety and Pharmacokinetics of Rhu-plasma Gelsolin in Hospitalized Subjects With CAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioAegis Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTI-201
Record Dates: First submitted 2018-03-02; First posted 2018-03-15 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Community-acquired Pneumonia
Keywords: Recombinant human plasma gelsolin (rhu-pGSN); Severe community-acquired pneumonia (sCAP); Adjunctive therapy
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: visibly indistinguishable therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single Dose 6 mg/kg (Experimental): Intravenous administration of recombinant human plasma gelsolin at 6 mg/kg v. placebo (NSS) in addition to standard of care
  Interventions: Drug: Recombinant Human Plasma Gelsolin; Other: Normal Saline Placebo
- Multiple Dose 6 mg/kg (Experimental): Intravenous administration of recombinant human plasma gelsolin at 6 mg/kg once per day for 3 days v. placebo (NSS) in addition to standard of care
  Interventions: Drug: Recombinant Human Plasma Gelsolin; Other: Normal Saline Placebo
- Multiple Dose 12 mg/kg (Experimental): Intravenous administration of recombinant human plasma gelsolin at 12 mg/kg once per day for 3 days v. placebo (NSS) in addition to standard of care
  Interventions: Drug: Recombinant Human Plasma Gelsolin; Other: Normal Saline Placebo
- Multiple Dose 24 mg/kg (Experimental): Intravenous administration of recombinant human plasma gelsolin at 24 mg/kg once per day for 3 days v. placebo (NSS) in addition to standard of care
  Interventions: Drug: Recombinant Human Plasma Gelsolin; Other: Normal Saline Placebo

INTERVENTIONS:
Drug: Recombinant Human Plasma Gelsolin — Recombinant human plasma gelsolin lyophilized for reconstitution, reconstituted in sterile water
  Other Names: rhu-pGSN
Other: Normal Saline Placebo — Normal saline in volume equivalent to drug
  Other Names: NSS (0.9% normal saline)

SUMMARY:
A Phase 1b/2a, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Recombinant Human Plasma gelsolin (rhu-pGSN) Added to Standard of Care in Subjects Hospitalized for Acute Community-acquired Pneumonia (CAP)

DETAILED DESCRIPTION:
A total of 32 patients hospitalized with CAP will be randomized sequentially into 4 ascending dosing levels. Each dosing cohort will include 8 subjects randomized 3:1 rhu-pGSN:placebo (6 rhu-pGSN subjects:2 placebo subjects). Patient, caregiver, and sponsor will be blinded to treatment. An unblinded pharmacist will prepare the infusion, but otherwise have no contact with subject.

Dose will be based on actual body weight. Dose escalation will involve 3 dose levels of rhu-pGSN (6, 12, and 24 mg/kg) in patients admitted for CAP. Dose escalation will only occur after post-therapy safety information on all subjects in the prior cohort has been reviewed at Day 7 for the single-dose [SD] and multiple-ascending dose [MAD] arms. The MAD portion of the study will commence once single doses of 6 mg/kg of rhu-pGSN are shown to be acceptably safe. The first 2 doses must be administered in the hospital, but the third dose can be given in a monitored outpatient setting where appropriate. Discharged subjects will return for follow-up 7 days after the initiation of therapy (Day 7) and on Day 28 for the End-of-Study Visit.

To assess safety and tolerability starting at the initiation of study therapy, subjects will undergo physical examinations (PE; including vital sign measurements), adverse event (AE) assessments, concomitant medication assessments, safety laboratory testing, and electrocardiograms (EKG) completed locally, and other testing as per local custom.

Once informed consent is obtained, the following procedures will be performed:

1. Randomize to currently enrolling treatment arm.
2. Perform PE and document radiographic evidence of pneumonia if not previously completed in preceding 36 hours; calculate Confusion, Urea >7 mmol/L, Respiratory rate ≥30/min, Blood pressure systolic <90 or diastolic ≤60, and age ≥65 years (CURB-65), Sequential Organ Failure Assessment (SOFA), and Pneumonia Severity Index (PSI) scores.
3. Obtain blood and sputum cultures, routine/standard labs, and EKG per standard of care (SOC) (if not already performed). The microbiology lab is encouraged to also perform sputum Gram-stains, antigen detection, immunoassay, and genomic diagnostic tests when available.
4. Draw blood for baseline pGSN levels, C-reactive protein (CRP), procalcitonin level, and 10 ml aliquot to be frozen for subsequent biomarker assays.

Screening laboratory and other tests can serve as baseline values for participants (no need to repeat lab tests at entry if done within the prior 36 hours unless dictated by SOC).

Obtain repeat chest x-rays (CXRs), computed tomography (CT) scans, and labs/cultures, etc. during the hospitalization if/when indicated by SOC.

Recalculate CURB-65 and ΔSOFA scores and redraw procalcitonin, pGSN, and biomarker samples on Day 3 or 4 and Day 7.

For the one dose in the SD arm and the first 2 doses in the multiple-dose arms, blood will be drawn within 30 minutes predose, immediately postdose, and 2, 8, 12 and/or 16, and 24 hours (± 30 minutes) after the end of infusion for analysis of plasma for maximum concentration (Cmax), time to maximum concentration (Tmax), terminal half-life (T1/2), area under the curve from time zero to 8 hours (AUC0-8), and area under the curve from time zero to infinity (AUCinf). Sampling at both the 12- and 16-hour time points is encouraged where feasible, but only one of these two times is required. Identical PK sampling is encouraged where feasible, but not required for the third (last) dose.

On Day 28, collect samples for analysis of pGSN levels and antibodies against pGSN.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained from subject
2. Domicile: home, assisted living, rehabilitation facility, or nursing home (as long as the prospective participant is capable of providing written informed consent)
3. Duration of infection precipitating hospitalization by history <14 days
4. Planned or actual admission to hospital with a primary diagnosis of CAP within 24 hours of presentation to the hospital
5. Primary admitting diagnosis of pneumonia supported by a compatible clinical presentation with a documented infiltrate consistent with pneumonia on chest radiograph or CT, as assessed by the admitting emergency-department (ED), clinic, or ward physician or equivalent caregiver

   * Recommended (not mandatory) guidance/discretionary criteria defining patients with CAP:

     * At least 2 symptoms: difficulty breathing, cough, production of purulent sputum, chest pain
     * At least 2 vital sign abnormalities: fever, tachycardia, tachypnea
     * At least one finding of other clinical signs and laboratory abnormalities: hypoxemia, clinical evidence of pulmonary consolidation, an elevated total white blood cell (WBC) count or leukopenia
     * Chest imaging showing new (or presumed new or worsening) infiltrates
   * Receipt of antibiotic treatment prior to presentation does not exclude the patient

Exclusion Criteria:

1. Pregnant or lactating women
2. Intubation, vasopressor support, or admission to the intensive care unit (ICU) directly from the ED/office (fluids for responsive hypotension is not a reason for exclusion)
3. Use of any investigational drug in the past 30 days
4. Hospitalization during the last 30 days
5. Residence within the last 30 days in long-term care facility where the patient remains persistently unable to participate in the routine activities of daily living
6. Active underlying cancer treated with systemic chemotherapy or radiation therapy during the last 30 days
7. Known or suspected immunosuppressive disease or therapy (including steroid use equivalent to prednisone ≥20 mg/day for >7 days or known advanced human immunodeficiency virus (HIV) infection with CD4 count ≤200/mm3; specific testing for HIV status or CD4 count is not required but can be done at the discretion of the caregivers)
8. Active congestive heart failure, myocardial infarction, or pulmonary embolism; cardiopulmonary arrest in last 30 days
9. Weight >100 kg
10. Otherwise unsuitable for study participation in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J DiNubile, MD, Study Chair — BioAegis Therapeutics Inc.
Locations (8):
- Australia (3):
  - Cairns Hospital, Cairns, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Footscray Hospital, Footscray, Victoria
- Georgia (5):
  - LTD Geo Hospitals, Mtskheta Multiprofile Medical Center, Mtskheta
  - JSC Rustavi Central Hospital, Rustavi
  - LTD Central University Clinic After Academic N. Kipshidze, Tbilisi
  - LTD S. Khechinashvili University Hospital, Tbilisi
  - LTD 5th Clinical Hospital, Tbilisi

REFERENCES:
- [Derived] Tannous A, Levinson SL, Bolognese J, Opal SM, DiNubile MJ. Safety and Pharmacokinetics of Recombinant Human Plasma Gelsolin in Patients Hospitalized for Nonsevere Community-Acquired Pneumonia. Antimicrob Agents Chemother. 2020 Sep 21;64(10):e00579-20. doi: 10.1128/AAC.00579-20. Print 2020 Sep 21. PMID 32690640

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 mg/kg Rhu-pGSN Single Dose: Intravenous administration of recombinant human plasma gelsolin at 6 mg/kg in addition to standard of care
- Placebo Single Dose: Intravenous administration of placebo (NSS) in addition to standard of care
- 6 mg/kg Rhu-pGSN Multiple Ascending Dose: Intravenous administration of recombinant human plasma gelsolin at 6 mg/kg in addition to standard of care once a day for 3 consecutive days
- 12 mg/kg Rhu-pGSN Multiple Ascending Dose: Intravenous administration of recombinant human plasma gelsolin at 12 mg/kg in addition to standard of care once a day for 3 consecutive days
- 24 mg/kg Rhu-pGSN Multiple Ascending Dose: Intravenous administration of recombinant human plasma gelsolin at 24 mg/kg in addition to standard of care once a day for 3 consecutive days
- Placebo Multiple Ascending Dose: Intravenous administration of placebo (NSS) in addition to standard of care once a day for 3 consecutive days
Period: Overall Study
Arm/Group | 6 mg/kg Rhu-pGSN Single Dose | Placebo Single Dose | 6 mg/kg Rhu-pGSN Multiple Ascending Dose | 12 mg/kg Rhu-pGSN Multiple Ascending Dose | 24 mg/kg Rhu-pGSN Multiple Ascending Dose | Placebo Multiple Ascending Dose
Started | 6 | 2 | 6 | 6 | 6 | 7
Completed | 5 | 2 | 6 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 mg/kg Rhu-pGSN Single Dose | Placebo Single Dose | 6 mg/kg Rhu-pGSN Multiple Ascending Dose | 12 mg/kg Rhu-pGSN Multiple Ascending Dose | 24 mg/kg Rhu-pGSN Multiple Ascending Dose | Placebo Multiple Ascending Dose | Total
Number analyzed (Participants) | 6 | 2 | 6 | 6 | 6 | 7 | 33
Age, Continuous [Mean (Full Range); unit: years] | 62.2 [35 to 81] | 64 [62 to 66] | 69.3 [56 to 83] | 55.3 [45 to 70] | 40 [22 to 66] | 64 [39 to 78] | 58.7 [22 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 5 | 3 | 4 | 3 | 17
  Male | 4 | 2 | 1 | 3 | 2 | 4 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 2 | 6 | 6 | 6 | 7 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  Georgia | 1 | 1 | 6 | 6 | 6 | 7 | 27
  Australia | 5 | 1 | 0 | 0 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment emergent adverse events were all adverse events (AEs) that occurred subsequent to enrollment. The seriousness of adverse events was judged by the site investigator.
Time Frame: 0-28 days
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg/kg Rhu-pGSN Single Dose | Placebo Single Dose | 6 mg/kg Rhu-pGSN Multiple Ascending Dose | 12 mg/kg Rhu-pGSN Multiple Ascending Dose | 24 mg/kg Rhu-pGSN Multiple Ascending Dose | Placebo Multiple Ascending Dose
Number analyzed (Participants) | 6 | 2 | 6 | 6 | 6 | 7
Participants
  Subjects with at least 1 TEAE | 4 | 2 | 4 | 3 | 2 | 4
  Subjects with at least 1 Serious TEAE | 1 | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Pharmacokinetics (PK) (Area Under the Rhu-pGSN Concentration - Time Curve)
Description: Determine AUC 0-t area under the plasma concentration-time curve of rhu-pGSN from 0-24 hours on dosing days (estimated by subtracting pre-injection concentrations from the measured concentrations at each time point). In the single-dose arm, the subject was given only 1 dose so that data from later days were not obtained. In the multiple-dose arms, samples were obtained for each of the 3 doses.
Time Frame: On Days 0-3, specimens were obtained just prior and immediately post dose and 2, 8,12 and/or 16 , and 24 hours post completion of IV administration. In the single-dose arm, only 1 dose was given and thus no data from later days were obtained.
Population: Results from participants given the 6 mg/kg rhu-pGSN dose included 4 subjects in the single-dose arm (samples from 1 subject were lost and 1 subject was withdrawn from the study) and from all 6 patients in the multiple-dose arm given this dose, yielding 10 patients for Dose 1. Only 6 patients were studied on Doses 2 and 3.
Measure: Mean (Standard Deviation); unit: µg*h/mL
Groups:
- 6 mg/kg Rhu-pGSN: Intravenous administration of recombinant human plasma gelsolin at 6 mg/kg in addition to standard of care (single dose and multiple doses once a day for 3 consecutive days)
- 12 mg/kg Rhu-pGSN: Intravenous administration of recombinant human plasma gelsolin at 12 mg/kg in addition to standard of care once a day for 3 consecutive days
- 24 mg/kg Rhu-pGSN: Intravenous administration of recombinant human plasma gelsolin at 24 mg/kg in addition to standard of care once a day for 3 consecutive days
Arm/Group | 6 mg/kg Rhu-pGSN | 12 mg/kg Rhu-pGSN | 24 mg/kg Rhu-pGSN
Number analyzed (Participants) | 10 | 6 | 6
µg*h/mL
  AUC 0-t, Day 1 | 984.4 (3798.3) | 3450.1 (586.5) | 6911.3 (1914.1)
  AUC 0-t, Day 2: number analyzed (Participants) | 6 | 6 | 6
  AUC 0-t, Day 2 | 674.3 (1062.4) | 2602.8 (755.3) | 1818.4 (4088.5)
  AUC 0-t, Day 3: number analyzed (Participants) | 6 | 6 | 6
  AUC 0-t, Day 3 | 447.4 (626.6) | 3081.8 (1283.5) | 4315.8 (3004.3)

3. Secondary Outcome: Pharmacokinetics (PK) (Maximum Observed Rhu-pGSN Plasma Concentration (Cmax))
Description: Maximum observed plasma concentration (Cmax) of rhu-pGSN in a 24 hours period after intravenous administration (estimated by subtracting pre-injection concentrations from the measured concentrations at each time point). For the 6 mg/kg dose, there were 4 evaluable subjects in the single-dose arm and 6 subjects in the multiple-dose arm at this dose, for a total of 10 evaluable subjects for Dose 1.
Time Frame: On Days 0-3, specimens were obtained just prior and immediately post dose and 2, 8, 12 and/or 16, and 24 hours post completion of IV administration. In the single-dose arm, only 1 dose was given and thus no data from later days were obtained.
Population: Results from participants given the 6 mg/kg rhu-pGSN dose included 4 subjects in the single-dose arm (samples from 1 subject were lost and 1 subject was withdrawn from the study) and from all 6 patients in the multiple-dose arm given this dose, yielding results from 10 patients for Dose 1.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | 6 mg/kg Rhu-pGSN | 12 mg/kg Rhu-pGSN | 24 mg/kg Rhu-pGSN
Number analyzed (Participants) | 10 | 6 | 6
µg/mL
  Cmax, Day 1 | 226.6 (393.3) | 291.9 (38.0) | 533.9 (139.9)
  Cmax, Day 2: number analyzed (Participants) | 6 | 6 | 6
  Cmax, Day 2 | 177.9 (128.4) | 292.0 (79.4) | 347.3 (274.7)
  Cmax, Day 3: number analyzed (Participants) | 6 | 6 | 6
  Cmax, Day 3 | 133.9 (86.0) | 320.6 (75.4) | 498.8 (275.3)

4. Other Pre Specified Outcome: Number of Participants With Anti-pGSN Antibodies (Immunogenicity) at the End of Study (Day 28)
Description: Number of participants who developed antibodies against pGSN at study day 28. Patients were first tested against less stringent screening criteria: if screen-positive, a stricter confirmatory test was performed; if screen-negative, no further immunogenicity testing was done.
Time Frame: Day 28
Population: In this analysis, participants receiving single or multiple doses are reported separately.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg/kg Rhu-pGSN Single Dose | Placebo Single Dose | 6 mg/kg Rhu-pGSN Multiple Ascending Dose | 12 mg/kg Rhu-pGSN Multiple Ascending Dose | 24 mg/kg Rhu-pGSN Multiple Ascending Dose | Placebo Multiple Ascending Dose
Number analyzed (Participants) | 2 | 2 | 6 | 6 | 6 | 6
Participants
  Screened, positive | 0 | 0 | 1 | 2 | 6 | 2
  Confirmed, positive | 0 | 0 | 1 | 0 | 2 | 0

5. Other Pre Specified Outcome: Baseline and Sequential Severity Scores
Description: CURB-65 (a 5 point score in which 1 point is allocated to the presence of each of the following: Confusion, Urea >7 mmol/L, Respiratory rate ≥30 breaths min, Blood pressure systolic <90 mmHg or diastolic ≤60 mmHg, and age ≥65 years); PSI (Pneumonia Severity Index, used to predict risk of morbidity and mortality and is classified in risk classes ranging from I to V from the lowest to highest risk as follows: Class I: PSI 0, class II: PSI 1-70, class III: PSI 71-90, class IV: PSI 91-130, class V: PSI >130); SOFA (Sequential Organ Failure Assessment, measured based on 6 variables each representing an organ system scored from 0 to 4 each (normal to severe organ dysfunction/failure), and reported as the sum (range 0-24))
Time Frame: Days 0-28
Population: Results are reported for the combined multiple rhu-pGSN vs. the placebo recipients with available data. One of the placebo recipients in the MAD phase died before dose completion. Since the changes were small across dosing groups, we combined the multi-dose arm in the analysis
Measure: Median (Full Range); unit: unitless
Groups:
- Combined Rhu-pGSN Multiple Ascending Dose: Intravenous administration of recombinant human plasma gelsolin at 6 mg/kg,12 mg/kg & 24mg/kg in addition to standard of care once a day for 3 consecutive days
- Combined Placebo Multiple Ascending Dose: Intravenous administration of placebo (NSS) in addition to standard of care once a day for 3 consecutive days
Arm/Group | Combined Rhu-pGSN Multiple Ascending Dose | Combined Placebo Multiple Ascending Dose | 6 mg/kg Rhu-pGSN Single Dose | Placebo Single Dose
Number analyzed (Participants) | 18 | 7 | 6 | 2
unitless
  CURB-65-Baseline | 0 [0 to 2] | 1 [0 to 2] | 1 [0 to 2] | 1 [1 to 1]
  Change in CURB-65 from Baseline to Day 28: number analyzed (Participants) | 18 | 6 | 4 | 2
  Change in CURB-65 from Baseline to Day 28 | 0 [-1 to 1] | 0 [-1 to 0] | 0 [-1 to 2] | -0.5 [-1 to 0]
  PSI score-Baseline: number analyzed (Participants) | 15 | 5 | 6 | 2
  PSI score-Baseline | 52 [38 to 91] | 78 [56 to 98] | 67.5 [46 to 119] | 69 [62 to 76]
  Change in PSI score from Baseline to Day 28: number analyzed (Participants) | 14 | 4 | 4 | 2
  Change in PSI score from Baseline to Day 28 | 0 [-10 to 1] | -5 [-10 to 0] | 0 [0 to 0] | 0 [0 to 0]
  SOFA score-Baseline | 1 [0 to 3] | 1 [0 to 4] | 1.5 [0 to 4] | 2 [2 to 2]
  Change in SOFA score from Baseline to Day 28: number analyzed (Participants) | 18 | 6 | 5 | 2
  Change in SOFA score from Baseline to Day 28 | -1 [-3 to 0] | -1 [-4 to 0] | -1 [-1 to 0] | -2 [-2 to -2]

ADVERSE EVENTS:
Time Frame: 0-28 days
Arm/Group | 6 mg/kg Rhu-pGSN Single Dose | Placebo Single Dose | 6 mg/kg Rhu-pGSN Multiple Ascending Dose | 12 mg/kg Rhu-pGSN Multiple Ascending Dose | 24 mg/kg Rhu-pGSN Multiple Ascending Dose | Placebo Multiple Ascending Dose
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/2 | 0/6 | 0/6 | 0/6 | 1/7
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/2 | 0/6 | 0/6 | 0/6 | 1/7
Other Adverse Events (participants affected / at risk) | 3/6 | 2/2 | 4/6 | 3/6 | 2/6 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 mg/kg Rhu-pGSN Single Dose (N=6) | Placebo Single Dose (N=2) | 6 mg/kg Rhu-pGSN Multiple Ascending Dose (N=6) | 12 mg/kg Rhu-pGSN Multiple Ascending Dose (N=6) | 24 mg/kg Rhu-pGSN Multiple Ascending Dose (N=6) | Placebo Multiple Ascending Dose (N=7)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 6 mg/kg Rhu-pGSN Single Dose (N=6) | Placebo Single Dose (N=2) | 6 mg/kg Rhu-pGSN Multiple Ascending Dose (N=6) | 12 mg/kg Rhu-pGSN Multiple Ascending Dose (N=6) | 24 mg/kg Rhu-pGSN Multiple Ascending Dose (N=6) | Placebo Multiple Ascending Dose (N=7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headaches (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03466073/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT03466073/SAP_001.pdf